CLINICAL TRIAL: NCT06071182
Title: Task-oriented Game Therapy Using Free Internet-videogame Enhances Upper Extremity Functions for Children With Cerebral Palsy: A Sham-controlled Study.
Brief Title: Task-oriented Game Therapy Using Enhances Functions in Children With Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mehmet.sonmez
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy
Keywords: Therapy; Rehabilitataion; Video game
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-oriented therapy (Experimental): Traditional physiotherapy for 30 minutes a day, twice a week for 4 weeks (Passive upper extremity Normal Joint Movements, 3-way and 1 set of 10 repetitions passive stretches for the shoulder (bilateral), 2-way, 1 set of 10 repetitions passive stretches at the elbow level) + 2 times a week a day Fruit ninja game on tablet in 20 minutes
  Interventions: Device: Task-oriented Fruit ninja game
- Sham-controlled (Sham Comparator): Same time traditional therapy + 5 minutes sham intervention
  Interventions: Other: sham-controlled therapy

INTERVENTIONS:
Device: Task-oriented Fruit ninja game — The fruit ninja game were played from tablet PC 20 minutes in a day and 2 times in a week for 4 weeks
  Arms: Task-oriented therapy
Other: sham-controlled therapy — The fruit ninja game playing video (https://www.youtube.com/watch?v=cAb0cAviA1s) was watched on the same tablet for 3 minutes a day, twice a week, for 4 weeks, and the wrist and wrist exercises were repeated for 2 minutes on a flat and smooth table. movements were made.
  Arms: Sham-controlled

SUMMARY:
Cerebral Palsy is an umbrella definition that refers to a disorder that occurs after a problem affecting a person's brain functions and has symptoms such as sensory, motor and mental deficits. Cerebral Palsy can cause serious functional losses in individuals. Various rehabilitation approaches have been developed and used to eliminate these functional losses. One of these approaches is a therapy technique called Task-oriented therapy, which focuses on completing tasks that mostly involve functional activities that the participating individuals do actively and repeatedly. There are various ways to perform task-oriented therapy. These can be achieved by motivating the individual to perform various tasks (cutting with scissors, buttoning, putting on and taking off legos, etc.) in an active, intense and repetitive manner, as well as through games played on devices such as tablet computers that have emerged with the developing technology. Thanks to their Android and touch features, such devices can motivate people to use their upper extremities functionally. Thanks to such applications, rehabilitation practices can be made more fun and effective results can be obtained. In the literature, it was seen that video game-based rehabilitation practices were used in individuals with cerebral palsy, but their effects on balance were mostly evaluated. Its effect on upper extremity functional capacity was mostly limited to feasibility studies. For these reasons, there is no data in the literature on this subject with quality results. The main purpose of this study is to determine whether upper extremity functional capacity can be improved by using the Tablet PC-based Fruit ninja game, which is easily accessible today, in the rehabilitation of individuals with cerebral palsy, using objective measurement tools.

DETAILED DESCRIPTION:
This study is a sham-controlled prospective non-invasive field study. A total of 22 participants were pre-registered for the study. However, when the inclusion criteria were applied, 4 participants whose GMFCS score was not between levels 1-3 but met other conditions were excluded from the study without taking preliminary measurements. A total of 18 participants were included in the study by taking preliminary measurements. Participants were randomly distributed (Computerized randomization (random.org)) into a nine-person study group and a placebo control group.

Traditional physiotherapy (Passive upper extremity Normal Joint Movements, 3-way and 1 set of 10 repetitions of passive stretching for the shoulder (bilateral), 2-directional and 1 set of 10 repetitions of passive stretching at the elbow level) was applied to the study group for 30 minutes a day, twice a week for 4 weeks, and then Fruit ninja game was played on the tablet for 20 minutes a day, twice a week.

The control group was treated with traditional physiotherapy (Passive upper extremity Normal Joint Movements, 3-way and 1 set of 10 repetitions passive stretching for the shoulder (bilateral), 2-way, 1 set of 10 repetitions passive stretching at the elbow level) for 30 minutes a day, twice a week for 4 weeks. For placebo purposes, the fruit ninja game playing video (https://www.youtube.com/watch?v=cAb0cAviA1s) was watched on the same tablet for 3 minutes a day, twice a week, for 4 weeks, and the movements in the game were repeated for 2 minutes on a flat and smooth table. Wrist movements were performed.

The first measurements of the participants participating in the study were taken after their last session the week before the study, as they came to rehabilitation twice a week, and their last measurements were taken after their last session in the 4th week and before their first session the following week. During this period, the participants' families were contacted to ensure that their children did not exercise or play any computer games at home. Measurements were carried out by the assistant researcher. Rehabilitation practices were carried out by the principal investigator and assistant investigator.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Cerebral Palsy with a doctor's report (Based on patient reports)
* Being between the ages of 6-18
* Having upper extremity involvement
* Being between levels 1-3 on the Expanded Gross Motor Function Classification (GMFS)
* Having the mental competence to understand the game being played

Exclusion Criteria:

* Those whose family did not sign a participation consent form

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Manual Dexterity | The change from baseline box and block test score at week 4
  Box and Block test is used. It is a measurement tool that measures gross comprehension skills. The number of cubes thrown one by one from one compartment to the other within 1 minute of a two-compartment box containing 150 cubes with dimensions of 2.5 cm*2.5 cm*2.5 cm is evaluated. It is done separately for right and left hands.
Hand function | The change from baseline nine hole peg test score at week 4
  Nine Hole Peg test is used It is a scale that evaluates participants functionally. It measures the time it takes to attach and remove 9 thin rods to a panel with 9 holes on it with the desired hand and return it to its box.
Grip strength | The change from baseline dinamometer score at week 4
  Analog dinamometer is used. Three times maximal grip strength is measured for both hands.
Range of movement | The change from baseline universal goniometer score at week 4
  Universal goniometers is used. Wrist flexion, wrist extension, radial and ulnar deviation scores (for both hands) are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet SÖNMEZ, MSc, Study Director — Erzurum Technical University
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No